CLINICAL TRIAL: NCT07304037
Title: The Effect of Skin-to-Skin Contact Applied in the Early Postpartum Period on Maternal Pain, Birth Satisfaction, and Maternal Vital Signs Dynamics
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Yasemin Dincel, Researcher Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2025/332
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Maternal Vital Signs; Skin-to-skin Contact; Birth Satisfaction
Keywords: maternal vital signs; skin-to-skin contact; birth satisfaction; Maternal outcomes; labor pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Immediately after birth, skin-to-skin contact is maintained continuously for one hour. Pain levels, birth satisfaction levels, and maternal vital signs (body temperature, oxygen saturation, heart rate, and blood pressure) are assessed at 30, 60, and 90 minutes postpartum.
  Interventions: Procedure: A solid hour of skin-to-skin contact
- Control Group (No Intervention): Following delivery, routine midwifery care is provided, and immediately after birth, at 30, 60, and 90 minutes, pain levels, satisfaction with the birth, and maternal physiological findings (body temperature, oxygen saturation, heart rate, and blood pressure) are assessed.

INTERVENTIONS:
Procedure: A solid hour of skin-to-skin contact — Immediately after birth, skin-to-skin contact is maintained for one hour without interruption. Pain levels, birth satisfaction levels, and maternal vital signs (body temperature, oxygen saturation, heart rate, and blood pressure) are assessed at 30, 60, and 90 minutes postpartum.
  Arms: Experimental Group

SUMMARY:
Skin-to-skin contact (STSC) initiated within the first hour after birth is a fundamental practice that supports both the mother's and the newborn's physiological and psychological adaptation (Çelik & Kök, 2022). The World Health Organization recommends at least 90 minutes of uninterrupted SKC immediately after birth and defines this practice as a mandatory component of care under the Baby-Friendly Hospital Initiative (World Health Organization, 2024; Abdulghani et al., 2018; Sharma, 2016). The positive effects of TTT on maintaining the newborn's temperature, glucose regulation, physiological stability, and mother-infant bonding have been proven (Sezici & Yiğit, 2020; Safar et al., 2018). In addition, it has been reported that it can shorten the third stage of labor by increasing maternal oxytocin release and reduce maternal stress and anxiety (Püsküllüoğlu et al., 2022; Harati Kabir et al., 2024).

In the study, mothers in the intervention group will receive one hour of uninterrupted TTT immediately after delivery; routine midwifery care will continue in the control group. In both groups, maternal pain levels, birth satisfaction, and vital signs (body temperature, oxygen saturation, heart rate, and blood pressure) will be assessed immediately after delivery, and at 30, 60, and 90 minutes.

The sample size was calculated using GPower, and a total of 68 participants (34 in each group) will be included in the study. Inclusion criteria include women aged 18 years or older who have had a full-term vaginal delivery and have a single, uncomplicated pregnancy. The data collection tools used will be the Demographic Information Form and the Visual Analog Scale (VAS).

The findings of the study are expected to enhance the quality of midwifery care by supporting the integration of TTT into clinical practice in early postpartum care.

DETAILED DESCRIPTION:
H1: There is a difference in pain scores measured using the Visual Analog Scale (VAS) between the group that received uninterrupted skin-to-skin contact for one hour after birth and the control group immediately after birth, at 30, 60, and 90 minutes.

H1: There is a difference in birth satisfaction scores measured using the Visual Analog Scale (VAS) between the group that received uninterrupted skin-to-skin contact for one hour after birth and the control group immediately after birth, at 30, 60, and 90 minutes.

H1: There is a difference between the group that received uninterrupted skin-to-skin contact for one hour after birth and the control group in terms of maternal body temperature, oxygen saturation, heart rate, and blood pressure measurements taken immediately after birth and at 30, 60, and 90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate in the study
* Be able to read, understand, and write in Turkish
* Be 18 years of age or older
* Have given birth vaginally
* Have given birth to a single baby
* Be at term (between 38-42 weeks of gestation)
* Have given birth vaginally in vertex presentation
* Estimated fetal weight between 2500-4000 grams
* Not having received any analgesia or anesthesia to relieve pain and fatigue during labor
* Having a pregnancy without maternal or fetal complications

Exclusion Criteria:

* Multiple pregnancies
* High-risk pregnancies with complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 68 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Visuel Analog Scale -Pain | At 30, 60, and 90 minutes after birth
  Min: 0- Max:10
Visuel Analog Scale- Birth satisfaction | At 30, 60, and 90 minutes after birth
  Min:0-Max:10

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Dinçel, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdulghani N, Edvardsson K, Amir LH. Worldwide prevalence of mother-infant skin-to-skin contact after vaginal birth: A systematic review. PLoS One. 2018 Oct 31;13(10):e0205696. doi: 10.1371/journal.pone.0205696. eCollection 2018. PMID 30379859
- [Result] Sharma A. Efficacy of early skin-to-skin contact on the rate of exclusive breastfeeding in term neonates: a randomized controlled trial. Afr Health Sci. 2016 Sep;16(3):790-797. doi: 10.4314/ahs.v16i3.20. PMID 27917213
- [Result] Safari K, Saeed AA, Hasan SS, Moghaddam-Banaem L. The effect of mother and newborn early skin-to-skin contact on initiation of breastfeeding, newborn temperature and duration of third stage of labor. Int Breastfeed J. 2018 Jul 16;13:32. doi: 10.1186/s13006-018-0174-9. eCollection 2018. PMID 30026787
- [Result] Kabir FH, Razavinia F, Keshavarz M, Mousavi SS, Haghani H. Effect of Companion Presence during Skin-to-Skin Contact on Maternal Anxiety: A Randomized Clinical Trial. Indian Pediatr. 2024 Mar 15;61(3):230-236. PMID 38469838
- [Result] Püsküllüoğlu, B., Göker, A. & Kosova, F. The effect of skin-to-skin contact on the expulsion time of the placenta and delivery hormones. DEU Tıp Dergisi, 2022, 36(3), 237-242. https://doi.org/10.18614/deutip1230581
- [Result] Sezici E, Yigit D. The Effect of Skin-to-Skin Contact on Maternal Anxiety, Heart Rate, and Oxygen Saturation during the Vaccination of One-Month-Old Infants. Compr Child Adolesc Nurs. 2020 Dec;43(4):410-420. doi: 10.1080/24694193.2020.1721614. Epub 2020 Feb 19. PMID 32073934
- [Result] Çelik, İ. & Kök, G. Examination of nurses' and midwives' knowledge and attitudes regarding early skin-to-skin contact between mother and newborn. Istanbul Development University Journal of Health Sciences, 2022, 17, 558-574.
- See also: World Health Organization, Skin-to-skin contact helps newborns breastfeed. World Health Organization. — https://www.who.int/westernpacific/newsroom/feature-stories/item/skin-to-skin-contact-helps-newborns-breastfeed